CLINICAL TRIAL: NCT07303413
Title: Approche Rythmique et Auditive Chez Les Enfants Avec Troubles du Spectre de l'Autisme (TSA)
Brief Title: A Rhythmic and Auditory Approach for Children With Autism Spectrum Disorders (ASD)
Acronym: THETABOOST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: IHU reConnect (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024-091_THETABOOST; 2025-A00707-42 (Other: ID-RCB)
Record Dates: First submitted 2025-06-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder
Keywords: language
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- short baseline (Experimental): First baseline of 4 weeks and a second baseline of 8 weeks
  Interventions: Behavioral: EEG recording; Behavioral: Picture recognition test
- medium baseline (Experimental): First baseline of 6 weeks and a second baseline of 6 weeks
  Interventions: Behavioral: EEG recording; Behavioral: Picture recognition test
- long baseline (Experimental): First baseline of 8 weeks and a second baseline of 4 weeks
  Interventions: Behavioral: EEG recording; Behavioral: Picture recognition test

INTERVENTIONS:
Behavioral: EEG recording — EEG recording while listening to natural sounds
Behavioral: Picture recognition test — Children will have 4 images in front of them and a sound recording will be played to tell them which image to choose. They will have to click on the one that corresponds to what was said in the sound recording.

SUMMARY:
The aim of this study is to assess the effectiveness of a rhythmic auditory training program in improving language skills in children with Autism Spectrum Disorder (ASD) who have a language acquisition disorder. The program focuses on training children to reproduce the syllable rhythms of speech, and the study will evaluate the children's language skills before and after participating in the program.

ELIGIBILITY:
Inclusion Criteria:

* aged between 3 and 6 at the time of inclusion
* Have received a formal medical diagnosis of ASD
* Have the consent of the parent(s)
* Declaration of a language delay by the parents
* Affiliated to social security or equivalent scheme

Exclusion Criteria:

* Conditions likely to interfere with the EEG and make its interpretation difficult, including severe epilepsy or cerebral malformations.
* Treatments likely to interfere with the EEG (sedatives, psychostimulants, anxiolytics, antidepressants).
* Known hearing impairment

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The difference in the progression of language acquisition measured by the difference in the number of images recognised in image recognition tests. | 12 weeks

SECONDARY OUTCOMES:
Comparison of Neural tracking of speech via EEG measurements of brain oscillatory activity before and after a session of listening to rhythmic sound. | 12 weeks
Comparison of theta/gamma frequency bands via EEG measurements of cerebral oscillatory activity before and after rhythmic auditory training | 12 weeks
Comparison of Phase Locking Value via EEG measurements of cerebral oscillatory activity before and after rhythmic auditory training | 12 weeks
Comparison of theta/gamma Phase-amplitude Coupling in auditory cortical areas via EEG measurements of cerebral oscillatory activity before and after rhythmic auditory training | 12 weeks
correlation between Neural tracking via EEG measurements of brain oscillatory activity during training and the language progression index. | 12 weeks
correlation between Phase Locking Value via EEG measurements of brain oscillatory activity during training and the language progression index. | 12 weeks
correlation between theta/gamma phase-amplitude coupling via EEG measurements of brain oscillatory activity during training and the language progression index. | 12 weeks
correlation between theta/gamma power via EEG measurements of brain oscillatory activity during training and the language progression index. | 12 weeks
correlation between Neural tracking via EEG measurements of brain oscillatory activity during training and the language progression index | 24 weeks
correlation between theta/gamma power via EEG measurements of brain oscillatory activity during training and the language progression index. | 24 weeks
correlation between theta/gamma phase-amplitude coupling via EEG measurements of brain oscillatory activity during training and the language progression index. | 24 weeks
correlation between Phase Locking Value via EEG measurements of brain oscillatory activity during training and the language progression index. | 24 weeks

IPD SHARING:
Plan to Share IPD: Undecided